CLINICAL TRIAL: NCT04180670
Title: Prevalence of Urinary Incontinence and Evaluation of Related Factors in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Prevalence of Urinary Incontinence and Evaluation of Related Factors in Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Meltem Uzun, Lecturer, Sanko University
Other Study IDs: Sanko
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Urinary Incontinence
Keywords: chronic Obstructive Pulmonary Disease; urinary incontinence; self-activity assesment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary incontinence (UI) is defined as involuntary urinary incontinence. In women with COPD, chronic coughing can often lead to UI. In this patient group, incontinence may be related to functional impairment, concomitant diseases and medications used. The aim of this study was to determine the incidence of urinary incontinence in patients with chronic obstructive pulmonary disease (COPD) and the factors that may be associated with urinary incontinence. The study included individuals who applied to the Pulmonary Diseases Policlinic of SANKO University Sani Konukoğlu Practice and Research Hospital and followed up with the diagnosis of COPD. The age, sex, height, weight, education level, smoking, exercise habits, fluid intake, medications and accompanying diseases such as heart disease, hypertension and diabetes will be recorded. Any prolapse or surgery will be questioned and noted. The disease severity will be determined by the forced expiratory volume (FEV1) value of the first second obtained from pulmonary function tests. Dyspnea score will also be determined by the Modified British Research Council (MBRC). Symptoms will be evaluated with the COPD Assessment Test (CAT). For urinary incontinence, the ICIQ-SF (International Urinary Incontinence Consultation) Questionnaire and Urinary Distress Inventory will be applied. In addition, the Leicester Cough Questionnaire will be used to assess your coughing functions, and the Activity-Self Assessment will be performed to determine the individual activity adequacy and the value of activities for individuals. All evaluations will be done only once with the help of the physiotherapist and asking the questions and recording the answers of the individual.

DETAILED DESCRIPTION:
rinary incontinence (UI) is defined as involuntary urinary incontinence. In women with COPD, chronic coughing can often lead to UI. In this patient group, incontinence may be related to functional impairment, concomitant diseases and medications used. The aim of this study was to determine the incidence of urinary incontinence in patients with chronic obstructive pulmonary disease (COPD) and the factors that may be associated with urinary incontinence. The study included individuals who applied to the Pulmonary Diseases Policlinic of SANKO University Sani Konukoğlu Practice and Research Hospital and followed up with the diagnosis of COPD. The age, sex, height, weight, education level, smoking, exercise habits, fluid intake, medications and accompanying diseases such as heart disease, hypertension and diabetes will be recorded. Any prolapse or surgery will be questioned and noted. The disease severity will be determined by the forced expiratory volume (FEV1) value of the first second obtained from pulmonary function tests. Dyspnea score will also be determined by the Modified British Research Council (MBRC). Symptoms will be evaluated with the COPD Assessment Test (CAT). For urinary incontinence, the ICIQ-SF (International Urinary Incontinence Consultation) Questionnaire and Urinary Distress Inventory will be applied. In addition, the Leicester Cough Questionnaire will be used to assess your coughing functions, and the Activity-Self Assessment will be performed to determine the individual activity adequacy and the value of activities for individuals. All evaluations will be done only once with the help of the physiotherapist and asking the questions and recording the answers of the individual.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD

Exclusion Criteria:

* 65 and above patients Patients with congenital anomalies that may cause incontinence Patients with neurological diagnosis that may cause incontinence
* Obese patients with BMI over 30
* Female patients with traumatic gynecological history
* Patients with incontinence after severe gynecological operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with COPD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
MMRC Dyspnea score | First day
  Grade shortness of breath that may occur during daily exercises. "0" means shortness of breath with heavy exercise and 5 means shortness of breath even when dressing and undressing.
COPD Assessment Test CAT | First day
  It is an eight-item short, easy-to-apply test that measures the effects of COPD and deterioration in health status. The change in two units or more at the individual patient level is clinically significant.
ICIQ-SF (International Urinary Incontinence Consultation) Survey | First day
  It consists of 6 questions. In the first two questions, the date of birth and gender are questioned, while in the third question the incidence of urinary incontinence is questioned in the fourth question. 5. Question "How much incontinence affects your daily life?" Is answered between 0 (does not affect it in any way) and 10 (very much affects) and makes you think that the quality of life gets worse as you get closer to 10. In question 6, the time of incontinence is questioned. The maximum value is 21. The higher the score, the lower the quality of life.
Urinary Distress Inventory | First day
  It consists of 6 questions and is graded as a four-point Likert. The first two questions address irritative symptoms (urgency, frequency, and pain), while questions 3 and 4 aim at stress symptoms, and the last two questions address obstructive or voiding symptoms.
Leicester Cough Survey | First day
  It consists of 19 items, three of which are physical, psychological and social. The items in the Leicester Cough Questionnaire were selected by clinical effect factor method. This method selects the subjects that the patients define as problems and differentiates them according to the importance of the patients. Topics are also divided into fields. The questionnaire is completed on a seven-point Likert Scale (1 = Always, 2 = Most of the time, 3 = Often, 4 = Sometimes, 5 = Occasionally, 6 = Rarely, 7 = Never). Higher scores indicate better health status. Total score; It is the sum of the scores of the three subheadings (physical, psychological and social).
Activity-Self Assessment | First day
  It is an individual-centered assessment tool consisting of 21 questions related to the individual's kendisi self alı related to the activity activity (how well it performs the activity) and value (how valuable / important the relevant activity is for itself). The first 11 questions are skills; 12.-16. questions between habits and 17.-21. items related to requests.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Uzun, PhD(c), Principal Investigator — Sanko University
Locations (1):
- SANKO University, Gaziantep, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided